CLINICAL TRIAL: NCT04260594
Title: Randomized, Open, Multicenter Study on the Efficacy and Safety of Arbidol Hydrochloride Tablets in Treating Pneumonia in Patients Infected With Novel Coronavirus (2019-ncov).
Brief Title: Clinical Study of Arbidol Hydrochloride Tablets in the Treatment of Pneumonia Caused by Novel Coronavirus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jieming QU (Other)
Responsible Party: Sponsor-Investigator, Jieming QU, professor, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Abdrcspc202001
Record Dates: First submitted 2020-02-06; First posted 2020-02-07 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: 2019-nCoV
MeSH Terms: interventions — umifenovir

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arbidol tablets + basic treatment (Experimental)
  Interventions: Drug: Arbidol; Other: basic treatment
- basic treatment (Sham Comparator)
  Interventions: Other: basic treatment

INTERVENTIONS:
Drug: Arbidol — Arbidol tablets: take 2 tablets/time, 3 times/day for 14-20 days
  Other Names: The basic treatment used by the investigator was based on the condition of the patient
  Arms: Arbidol tablets + basic treatment
Other: basic treatment — basic treatment

SUMMARY:
In the absence of 2019-ncov specific therapeutic drugs, arbidol is effective against a variety of coronaviruses in vitro pharmacodynamics. In order to observe the efficacy and safety of arbidol in the treatment of 2019-ncov infected pneumonia, this study is planned.

DETAILED DESCRIPTION:
In December 2019, Wuhan, in Hubei province, China, became the center of an outbreak of pneumonia of unknown cause. In a short time, Chinese scientists had shared the genome information of a novel coronavirus (2019-nCoV) from these pneumonia patients and developed a real-time reverse transcription PCR (real time RT-PCR) diagnostic assay. The number of cases of infection with 2019-nCoV identified in Wuhan increased markedly over the later part of January 2020, with cases identified in multiple other Provinces of China and internationally. Mathematical models of the expansion phase of the epidemic suggested that sustained person-to-person transmission is occurring, and the R-zero is substantially above 1, the level required for a self-sustaining epidemic in human populations.

There is currently no specific treatment for 2019-ncov-infected pneumonia. Arbidol tablet is a non-nucleoside broad-spectrum antiviral drug with immune-enhancing effect. Abidor is pharmacodynamic in vitro against a variety of coronaviruses.This is a randomized, open, multicenter clinical study of pneumonic subjects diagnosed with 2019-ncov infection. The main objective was to compare the viral negative conversion rate in the first week after the subjects were randomized to arbidol plus basic treatment.

In this study, 380 eligible patients with pneumonia diagnosed with 2019-ncov infection were randomly assigned to one of two treatment groups at a 1:1 ratio.

patients will receive one of two treatment regimens: A .Abidor tablets + basic treatment B. basic treatment Arbidol tablets: take 2 tablets/time, 3 times/day for 14-20 days Basic treatment :The basic treatment used by the investigator was based on the condition of the patient.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 to 65 years old (including 18 and 65 years);
2. male and non-pregnant female;
3. respiratory tract specimens or hematology samples detected positive results of SARS-CoV-2 by real-time transcriptase polymerase chain reaction (RT-PCR).
4. mild clinical status, defined as having mild clinical symptoms but no signs of pneumonia on imaging or moderate clinical status, defined as having fever, respiratory symptoms and pneumonia on imaging or severe clinical status, defined as having an oxygen saturation (SaO2) of 93% or less at ambient air or a ratio of the partial pressure of oxygen (PaO2) to the fraction of inspired oxygen (FiO2) at or below 400 mgHg, which can be rectified by oxygen inhalation through nasal catheter or face mask.

Exclusion Criteria:

included a physician decision that involvement in the trial was not in the patient's best interest, known allergic reaction and / or severe allergic to arbidol, blood system dysfunction (platelet count <100×109/L, hemoglobin level <90g/L), severe liver dysfunction (total bilirubin level >2 times the normal upper limit, aspartic aminotransferase and alanine aminotransferase levels >3 times normal upper limit),severe renal dysfunction (serum creatinine >1.5 times the upper limit of normal value, calculated creatinine clearance rate <50 ml/min), treated with arbidol before admission, history of severe heart disease or clinically significant arrhythmia considered unsafe for the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2020-02-08 (Actual); Primary Completion 2020-03-12 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Virus negative conversion rate in the first week | first week

SECONDARY OUTCOMES:
Virus negative conversion rate | 14-20 days
  virus negative conversion rate in second week, overall virus negative conversion rate
Antipyretic rate | 14-20 days
  defined as: the rate of Axillary temperature ≤37.5 ℃ for at least 48h
Symptom relief time | 14-20 days
  time to relieve symptoms of fever, cough, dyspnea, myalgia, etc
Finger oxygen improvement rate | 14-20 days
  no adjuvant oxygen therapy, resting oxygen saturation>95%, oxygenation index>350
Disease progression rate | 14-20 days
  Mild, common type progression to severe or critical illness rate
Mortality rate | 14-20 days
Incidence of severe adverse reactions | 14-20 days
Change curve of peripheral blood lymphocyte count | 14-20 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Medical School of Shanghai Jiaotong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao J, Zhang J, Jin Y, Tang Z, Hu K, Sun H, Shi M, Yang Q, Gu P, Guo H, Li Q, Zhang H, Li C, Yang M, Xiong N, Dong X, Xu J, Lin F, Wang T, Yang C, Huang B, Zhang J, Chen S, He Q, Zhou M, Qu J. A trial of arbidol hydrochloride in adults with COVID-19. Chin Med J (Engl). 2022 Jul 14;135(13):1531-8. doi: 10.1097/CM9.0000000000002104. Online ahead of print. PMID 35830201